CLINICAL TRIAL: NCT02585843
Title: Pilot Study of Natriuretic Versus Standard Doses of Mineralocorticoid Receptor Antagonists in Heart Failure and Loop Diuretic Resistance in Outpatients
Brief Title: Mineralocorticoid Receptor Antagonists (MRA) in Heart Failure (HF) and Loop Diuretic Resistance
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Arthur R. Garan, Assistant Professor of Medicine at the Columbia University Medic, Dept of Medicine Cardiology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AAAO9102
Record Dates: First submitted 2015-08-30; First posted 2015-10-23 (Estimated); Results first posted 2019-07-23 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-07

CONDITIONS: Heart Failure
Keywords: Heart Failure; Mineralocorticoid receptor antagonists; Loop diuretic resistance
MeSH Terms: conditions — Heart Failure | interventions — Canrenoic Acid; Spironolactone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- High-dose (Experimental): Spironolactone 100mg: 100mg/day of spironolactone (2 capsules), PO (oral) for 7 days
  Interventions: Drug: Spironolactone 100mg
- Standard of Care (Active Comparator): Spironolactone 25mg: 25mg/day of spironolactone, PO (oral)
  Interventions: Drug: Spironolactone 25mg

INTERVENTIONS:
Drug: Spironolactone 100mg — 2 capsules of study medication consist of 100mg, PO (oral) for 7 days
  Other Names: Aldactone
  Arms: High-dose
Drug: Spironolactone 25mg — 25mg/day of spironolactone
  Other Names: Aldactone
  Arms: Standard of Care

SUMMARY:
This is a prospective, single-center, double-blind and randomized placebo controlled trial for evaluation of a 7-day 100mg daily dose of spironolactone on weight loss and resolution of signs and symptoms of congestion in outpatients with acute decompensated heart failure (ADHF). Patients who are not responding to their current loop diuretics will be considered for this study. Mineralocorticoid receptor antagonists (MRAs) are recommended as standard of care in management of heart failure (HF) patients. However, recommended doses of MRAs (spironolactone 25mg/daily or eplerenone 50mg/daily) will not have any impact on signs and symptoms of volume overload. Therefore, the proposed study will aim to show the impact of this outpatient regimen to improve diuresis and possible reduction in hospitalization for further diuretic management in HF patients with signs and symptoms of congestion.

DETAILED DESCRIPTION:
The incidence and prevalence of heart failure (HF) is rising with more than 5 million Americans suffering from this syndrome. Hospitalization rates for acute decompensated heart failure (ADHF) are also remarkably high, exceeding more than 1 million admissions per year. Congestion is the main cause of hospitalization for ADHF. Loop diuretics as the main therapy for decongestion, often are not adequate since many patients with ADHF develop "loop diuretic resistance". These patients will require hospitalization for intravenous diuretic or other advanced decongestion therapies. Thus, novel decongestion therapies are needed to decrease hospital admission rates and subsequent complications of multiple hospitalizations. Hyperaldosteronism, not only is a pivotal pathogenic factor in HF, but also contributes to loop diuretic resistance. Attempts for normalization of circulatory aldosterone with mineralocorticoid receptor antagonists (MRAs), mainly spironolactone, have shown to decrease mortality in HF patients with reduced left ventricular ejection fraction (LVEF). Moreover, MRAs significantly decrease the rate of rehospitalization in both HF with preserved and reduced LVEF. The dose of spironolactone in these trials is 25mg daily. However, this dose does not increase natriuresis (urinary sodium excretion). Natriuresis is achieved with higher doses of MRAs. Therefore, the primary aim of this study is to examine the efficacy of 7-day 100mg daily of spironolactone on weight loss and resolution of signs and symptoms of congestion in patients aged 60 years with ADHF and loop diuretic resistance.

ELIGIBILITY:
Inclusion Criteria:

* History of heart failure with either reduced or preserved ejection fraction for 3 months
* Patients with New York Heart Association (NYHA) class II- IV heart failure symptoms, with at least one worsening symptom (Dyspnea on exertion, shortness of breath, orthopnea, early satiety) and one sign of congestion (pulmonary rales, elevated jugular venous pressure10cmHg, peripheral edema and ascites)
* Decision by primary cardiologist or heart failure (HF) specialist to increase the home diuretic dose
* Stable treatment with beta-blockers for 1 month unless contraindicated (i.e. intolerance, bradycardia) as specified by primary cardiologist/HF provider
* Stable treatment with angiotensin converting enzyme-1 (ACE-1) or angiotensin receptor blocker (ARB) for 1 month
* Spironolactone dose 25mg or eplerenone 50mg per day
* Daily furosemide or furosemide equivalent dose of 80mg or greater
* Serum potassium concentration 4.5 mmol/L or 5.0 mmol/L if on potassium supplements
* Estimated Glomerular Filtration Rate (eGFR) by Modification of Diet in Renal Disease (MDRD) equation 40 ml/min/1.73

Exclusion Criteria:

* Inability to complete informed consent form
* Allergy or intolerance to spironolactone
* Systolic blood pressure <100 mmHg
* Patient in need of hospitalization per cardiologist decision
* Current inotrope dependency
* Current mechanical circulatory support
* Acute coronary syndromes or unstable angina within the past 4 weeks
* History of cardiac transplant
* Obstructive cardiac valvular disease
* Primary hypertrophic cardiomyopathy, infiltrative cardiomyopathy
* Significant ventricular arrhythmia necessitating defibrillator therapy within the past 14 days
* Atrioventricular conduction abnormality greater than first-degree block
* Primary liver disease resulted in cirrhosis or abnormal liver function tests (transaminases and alkaline phosphatase levels 3 times the upper limit of normal
* Acute malignancy
* Active infection requiring antimicrobial treatment (Suppression antimicrobial for chronic infections are exempt)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arthur R Garan, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | High-dose | Standard of Care
Started | 10 | 10
Completed | 9 | 10
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High-dose | Standard of Care | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (9) | 63.5 (15) | 62.6 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 4 | 5 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: African American | 4 | 2 | 6
  Race/Ethnicity: Hispanic | 5 | 8 | 13
  Race/Ethnicity: White | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20
Baseline 6 minute walk test [Mean (Standard Deviation); unit: meters] | 177 (78) | 196 (68) | 187 (69)

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Weight
Description: change in body weight measured in kilograms between weight at baseline and weight at 7 days
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: kilogram
Arm/Group | High-dose | Standard of Care
Number analyzed (Participants) | 9 | 10
kilogram | -1.9 (2.0) | -1.9 (1.1)

2. Secondary Outcome: Change in Estimated Jugular Venous Pressure (cmH2O)
Description: Change in estimated jugular venous pressure by physical exam in cmH2O between baseline and 7 days
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: cmH2O
Arm/Group | High-dose | Standard of Care
Number analyzed (Participants) | 9 | 10
cmH2O | -3.2 (2.5) | -3.9 (2.2)

3. Secondary Outcome: Change in 6-minute Walk Test Distance (6MWT)
Description: At baseline and final visit. The 6MWT will be conducted per American Thoracic Society guidelines.
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | High-dose | Standard of Care
Number analyzed (Participants) | 9 | 10
meters | 36 (46) | 36 (41)

4. Secondary Outcome: Change in Score on the Visual Analogue Scale (VAS)
Description: Dyspnea will be assessed at baseline and at 7 days with the score on the visual analogue scale (VAS). The scores range from 0 (minimum) to 100 (maximum) with higher numbers representing improvements in dyspnea (i.e. better) and lower numbers representing worsening of dyspnea (i.e. worse).
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High-dose | Standard of Care
Number analyzed (Participants) | 9 | 10
units on a scale | 26 (34) | 25 (17)

5. Secondary Outcome: Change From Baseline to Day 7 on the Seven-Level Likert Scale
Description: Dyspnea will be assessed using a Seven-Level Likert Scale at baseline and the day 7 visit. The outcome measure will be reported as a difference between these two assessments (value at 7 days minus the value at baseline). The values on this scale range from 1 to 7 with higher numbers indicating overall better subjective assessment related to the symptom of dyspnea. Therefore, positive numbers represent an overall improvement in dyspnea during the study intervention and the higher (more positive) this difference is, the better the subject's relief of dyspnea at the conclusion of the study intervention.
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High-dose | Standard of Care
Number analyzed (Participants) | 9 | 10
units on a scale | 2.1 (0.9) | 2.6 (0.5)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | High-dose | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 1/10 | 0/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High-dose (N=10) | Standard of Care (N=10)
Hyperkalemia (Renal and urinary disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-08-30): https://cdn.clinicaltrials.gov/large-docs/43/NCT02585843/Prot_000.pdf
  • Statistical Analysis Plan (2015-08-30): https://cdn.clinicaltrials.gov/large-docs/43/NCT02585843/SAP_001.pdf